CLINICAL TRIAL: NCT06186869
Title: Effects of Two Different Exercise Programs Combined With the Mediterranean Diet on Inflammatory Status in Subjects With Obesity and NAFLD
Brief Title: Effects of Two Different Exercise Programs and Diet in Obese Subjects With NAFLD
Acronym: Obesity_AF
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Azienda Ospedaliera Specializzata in Gastroenterologia Saverio de Bellis (Other)
Collaborators: Antonella Bianco (Unknown); Isabella Franco (Unknown)
Responsible Party: Principal Investigator, Dr. Endrit Shahini, Dr, Azienda Ospedaliera Specializzata in Gastroenterologia Saverio de Bellis
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AF_001
Record Dates: First submitted 2023-11-09; First posted 2024-01-02 (Actual); Last update posted 2025-05-01 (Actual); Status verified 2025-04

CONDITIONS: Obesity; NAFLD
Keywords: Obesity; Physical Exercise; systemic inflammation; NAFLD
MeSH Terms: conditions — Obesity; Non-alcoholic Fatty Liver Disease; Motor Activity | interventions — Exercise; Diet

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Aerobic Exercise and Mediterranean Diet (Active Comparator): Subjects randomized and assigned to this intervention group will follow the low glycaemic index Mediterranean diet and simultaneously perform 180 minutes of moderate-intensity aerobic exercise per week for 4 months. Intervention type: aerobic exercise and Mediterranean diet.
  Interventions: Behavioral: Aerobic Exercise and diet intervention
- HITT and Mediterranean Diet (Active Comparator): Subjects randomized and assigned to this intervention group will follow the low glycaemic index Mediterranean diet and simultaneously perform 150 minutes per week of high-intensity interval exercise (HITT) in the gym for 4 months. Intervention type: HIIT and Mediterranean diet.
  Interventions: Behavioral: Hiit and diet intervention
- Mediterranean Diet (Active Comparator): Subjects randomized and assigned to this intervention group will follow the low-glycaemic index Mediterranean diet for 4 months. Intervention type: Mediterranean Diet.
  Interventions: Behavioral: Diet

INTERVENTIONS:
Behavioral: Aerobic Exercise and diet intervention — subjects randomized and assigned to one intervention group, will follow the low glycaemic index Mediterranean diet and simultaneously perform moderate-intensity aerobic exercises
  Arms: Aerobic Exercise and Mediterranean Diet
Behavioral: Hiit and diet intervention — subjects randomised and assigned to one intervention group, will follow the low glycaemic index Mediterranean diet and simultaneously perform high-intensity interval exercises in the gym
  Arms: HITT and Mediterranean Diet
Behavioral: Diet — subjects randomised and assigned to this intervention group will follow the low-glycaemic index Mediterranean diet
  Arms: Mediterranean Diet

SUMMARY:
The aim of the study is to estimate the effectiveness of two different exercise programs combined with the Mediterranean diet versus diet alone on inflammatory status in subjects aged 18-65 years with obesity (BMI>30) and Non-Alcoholic Fatty Liver Disease (NAFLD) (CAP >248 dB/m).

DETAILED DESCRIPTION:
The main objective of the study is to estimate the effect of two exercise programs of different type and intensity combined with a Low Glycaemic Index Mediterranean Diet (LGIMD) compared to diet alone on the systemic inflammation index (SII) and biomarkers related to the inflammatory state: TNF-alpha; IL-1, IL-6, IL-10, CK-18, PCR and VES, in patients with obesity and NAFLD aged 18-65 years after a 4-month intervention.

The secondary objectives are: to assess whether the adoption of the two exercise programs of different types and intensities associated with an LGIMD compared to diet alone in patients with obesity and NAFLD can significantly modify body composition, inhibiting the risk of sarcopenia, in turn, favored by NAFLD, improve physical efficiency (fitness), understood as cardio-respiratory fitness muscular strength and flexibility, may also lead to improvements regarding the gut microbiota, in terms of abundance of microbial taxa, by studying, starting from the data obtained from the 16S, the metabolic pathways of the microbiota and fecal metabolome, as well as Quality of Life, by filling in specific questionnaires, and the evaluation of the fatty acid profile of erythrocyte membranes.

The two different types of exercise will be: - outdoor walking, understood as a moderate-intensity aerobic exercise, carried out 4 times a week, for a duration of 60 minutes for 4 months; - High-Intensity Interval Training carried out 3 times a week, for a period of 50 minutes at a time for 4 months in a gymnasium affiliated with the organization.

The diet will be the same for all project participants and will follow advice based on the Low Glycaemic Index Mediterranean Diet. All subjects will be followed by specialized personnel regarding both diet and exercise.

ELIGIBILITY:
Inclusion Criteria:

* BMI ≥ 30 kg/m2 or an abdominal circumference (waist) > 94 cm in men and > 80 cm in women (IDF criteria for the definition of abdominal obesity) with or without the characteristics that characterise metabolic syndrome
* Age range 18-65 years, both sexes
* Diagnosis of hepatic steatosis, formulated on the basis of recognised criteria (fibroscan (CAP (controlled attenuation parameter) > 238 dB/m)).

Exclusion Criteria:

* Normal and underweight subjects
* Presence of any pathology that may influence the presence of steatosis apart from pathologies that are inclusion criteria, neurological and psychiatric pathologies, gastrointestinal, oncological and cardiovascular diseases
* Pregnancy or breastfeeding
* Subjects with osteoarticular pathologies that may prevent regular exercise
* Inability to quantify the degree of NAFLD by Fibroscan
* Person not in possession of a medical certificate of fitness for non-competitive physical activity.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2023-10-02 (Actual); Primary Completion 2025-12-15 (Estimated); Study Completion 2026-12-23 (Estimated)

PRIMARY OUTCOMES:
The effect of diet and exercise on systemic inflammatory status | at baseline and day120
  To estimate the effect of two exercise programs of different types and intensity combined with a Mediterranean Low Glycaemic Index Diet (LGIMD) compared to diet alone on the systemic inflammation index (SII) and biomarkers related to the inflammatory state:
  C-reactive protein (CRP) and Erythrocyte sedimentation rate (ESR) were measured after venous blood sampling.
  Proinflammatory (TNF-alpha; IL-1, IL-6, CK-18) and anti-inflammatory (IL-10) cytokines will be measured using commercially available ELISA tests for each.

SECONDARY OUTCOMES:
The effect of diet and exercise on body composition | At baseline, day 60, and day 120
  To evaluate whether adopting two exercise programs of different types and intensities combined with an LGIMD versus diet alone in patients with obesity and NAFLD can significantly change body composition assessed by BIA and anthropometric data measurement.
The effect of diet and exercise on the gut microbiota | At baseline and day 120
  To investigate in patients with obesity and NAFLD, whether the adoption of the two programmes of Exercise of different types and intensities associated with an LGIMD compared to diet alone can improve the gut microbiota, in terms of abundances of microbial taxa, by studying, from the data obtained from the 16S, the metabolic pathways of the microbiota and faecal metabolome.
The effect of diet and exercise on quality of life | At baseline and day 120
  To evaluate the improvements in Quality of Life, by filling out specific questionnaires, following the adoption of the two programmes of Exercise of different types and intensities combined with an LGIMD versus diet alone in patients with obesity and NAFLD for 4 months.
  The questionnaire is divided into 8 domains, and each of the 8 summed scores is transformed linearly on a scale from 0 (negative health) to 100 (positive health) to provide a score for each subscale. Each subscale can be used independently. Scores < 50 indicate negative health, and > 51 indicate positive health.
The effect of diet and exercise on the fatty acid profile of erythrocyte membranes | At baseline and day 120
  All human blood samples will be treated with chloroform: methanol (2:1, v/v) and centrifuged. The lower layer, containing fatty acids, will be removed with care, replaced in a new tube, and dried by a centrifugal evaporator. The fatty acid methyl ester (FAME) will be obtained by adding toluene and BF3. Samples will be collected, transferred into a vial, and analyzed by gas chromatography.
The effect of diet and exercise on the risk of sarcopenia | At baseline and day 120
  To evaluate whether the adoption of two exercise programmes of different types and intensities combined with an LGIMD versus diet alone in patients with obesity and NAFLD can reduce the risk of sarcopenia closely related to NAFLD as assessed by measuring muscle mass (via BIA), muscle strength (handgrip test) and physical performance (SHORT PHYSICAL PERFORMANCE BATTERY (SPPB)).
The effect of diet and exercise on the peptides of Integrity Intestinal Barrier | At baseline and day 120
  Zonulin, I-FABP, DAO, and D-lactate assays will be performed using commercially available ELISA assays for each peptide.
The effect of diet and exercise on the Intestinal dysbiosis | At baseline and day 120
  The intestinal dysbiosis will be evaluated by assaying Indole using a colorimetric analytical method as a marker of fermentative dysbiosis, Skatole, a marker of putrefactive dysbiosis, will be assessed using a refined chromatographic method with fluorimetric detection. Both assays will be conducted on a urine sample.

CONTACTS AND LOCATIONS:
Overall Officials: Endrit Shahini, MD, Principal Investigator — IRCCS Saverio de Bellis
Locations (1):
- IRCCS De Bellis, Castellana Grotte, Bari, Italy

REFERENCES:
- [Background] Ye Q, Zou B, Yeo YH, Li J, Huang DQ, Wu Y, Yang H, Liu C, Kam LY, Tan XXE, Chien N, Trinh S, Henry L, Stave CD, Hosaka T, Cheung RC, Nguyen MH. Global prevalence, incidence, and outcomes of non-obese or lean non-alcoholic fatty liver disease: a systematic review and meta-analysis. Lancet Gastroenterol Hepatol. 2020 Aug;5(8):739-752. doi: 10.1016/S2468-1253(20)30077-7. Epub 2020 May 12. PMID 32413340
- [Background] Miryan M, Darbandi M, Moradi M, Najafi F, Soleimani D, Pasdar Y. Relationship between the Mediterranean diet and risk of hepatic fibrosis in patients with non-alcoholic fatty liver disease: A cross-sectional analysis of the RaNCD cohort. Front Nutr. 2023 Feb 22;10:1062008. doi: 10.3389/fnut.2023.1062008. eCollection 2023. PMID 36908910
- [Background] Sanyal AJ, Anstee QM, Trauner M, Lawitz EJ, Abdelmalek MF, Ding D, Han L, Jia C, Huss RS, Chung C, Wong VW, Okanoue T, Romero-Gomez M, Muir AJ, Afdhal NH, Bosch J, Goodman Z, Harrison SA, Younossi ZM, Myers RP. Cirrhosis regression is associated with improved clinical outcomes in patients with nonalcoholic steatohepatitis. Hepatology. 2022 May;75(5):1235-1246. doi: 10.1002/hep.32204. Epub 2022 Feb 7. PMID 34662449
- [Background] Misciagna G, Del Pilar Diaz M, Caramia DV, Bonfiglio C, Franco I, Noviello MR, Chiloiro M, Abbrescia DI, Mirizzi A, Tanzi M, Caruso MG, Correale M, Reddavide R, Inguaggiato R, Cisternino AM, Osella AR. Effect of a Low Glycemic Index Mediterranean Diet on Non-Alcoholic Fatty Liver Disease. A Randomized Controlled Clinici Trial. J Nutr Health Aging. 2017;21(4):404-412. doi: 10.1007/s12603-016-0809-8. PMID 28346567
- [Background] Franco I, Bianco A, Diaz MDP, Bonfiglio C, Chiloiro M, Pou SA, Becaria Coquet J, Mirizzi A, Nitti A, Campanella A, Leone CM, Caruso MG, Correale M, Osella AR. Effectiveness of two physical activity programs on non-alcoholic fatty liver disease. a randomized controlled clinical trial. Rev Fac Cien Med Univ Nac Cordoba. 2019 Feb 27;76(1):26-36. doi: 10.31053/1853.0605.v76.n1.21638. PMID 30882339
- [Background] Franco I, Bianco A, Mirizzi A, Campanella A, Bonfiglio C, Sorino P, Notarnicola M, Tutino V, Cozzolongo R, Giannuzzi V, Aballay LR, Buongiorno C, Bruno I, Osella AR. Physical Activity and Low Glycemic Index Mediterranean Diet: Main and Modification Effects on NAFLD Score. Results from a Randomized Clinical Trial. Nutrients. 2020 Dec 28;13(1):66. doi: 10.3390/nu13010066. PMID 33379253
- [Background] Calabrese FM, Disciglio V, Franco I, Sorino P, Bonfiglio C, Bianco A, Campanella A, Lippolis T, Pesole PL, Polignano M, Vacca M, Caponio GR, Giannelli G, De Angelis M, Osella AR. A Low Glycemic Index Mediterranean Diet Combined with Aerobic Physical Activity Rearranges the Gut Microbiota Signature in NAFLD Patients. Nutrients. 2022 Apr 23;14(9):1773. doi: 10.3390/nu14091773. PMID 35565740
- [Background] Bianco A, Franco I, Curci R, Bonfiglio C, Campanella A, Mirizzi A, Fucilli F, Di Giovanni G, Giampaolo N, Pesole PL, Osella AR. Diet and Exercise Exert a Differential Effect on Glucose Metabolism Markers According to the Degree of NAFLD Severity. Nutrients. 2023 May 10;15(10):2252. doi: 10.3390/nu15102252. PMID 37242135
- [Background] Xu M, Chen R, Liu L, Liu X, Hou J, Liao J, Zhang P, Huang J, Lu L, Chen L, Fan M, Chen X, Zhu X, Liu B, Hu P. Systemic immune-inflammation index and incident cardiovascular diseases among middle-aged and elderly Chinese adults: The Dongfeng-Tongji cohort study. Atherosclerosis. 2021 Apr;323:20-29. doi: 10.1016/j.atherosclerosis.2021.02.012. Epub 2021 Feb 20. PMID 33773161